CLINICAL TRIAL: NCT04915729
Title: A Phase III Multi-centre, Prospective, Randomised, Open Label, Blinded Endpoint (PROBE), Active-controlled Parallel Group Trial to Assess Efficacy and Safety of Tenecteplase Versus Alteplase in Chinese Patients With Acute Ischaemic Stroke Within 4.5 Hours After Stroke Onset
Brief Title: A Study in Chinese Patients to Compare How Tenecteplase and Alteplase Given After a Stroke Improve Recovering of Physical Activity
Acronym: ORIGINAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1123-0040
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase treatment group (Experimental): Chinese patients with AIS were screened (visit 1) and randomised (visit 2a) when admitted. Patients received a single dose of tenecteplase, 0.25 mg/kg via intravenous (iv) bolus no later than 4.5 hours (h) after symptom onset. Visits on Day 1 consisted of two further visits (Visit 2b and Visit 2c) that were performed 1 h and 2 h after the start of the treatment. Visits 3 to 5 for continuous follow-up were performed on day 2, 8 and 30 after the start of the treatment. Treated patient performed a 90-day follow-up visit after the treatment to complete the study.
  Interventions: Drug: tenecteplase
- Alteplase active control group (Active Comparator): Chinese patients with AIS were screened (visit 1) and randomised (visit 2a) when admitted. Patients received a single dose of alteplase, 0.9 mg/kg, 10% via intravenous (iv) bolus and the remaining 90% of the total dose administered as an iv infusion over 1 h no later than 4.5 hours (h) after symptom onset. Visits on Day 1 consisted of two further visits (Visit 2b and Visit 2c) that were performed 1 h and 2 h after the start of the treatment. Visits 3 to 5 for continuous follow-up were performed on day 2, 8 and 30 after the start of the treatment. Treated patient performed a 90-day follow-up visit after the treatment to complete the study.
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: tenecteplase — tenecteplase
  Arms: Tenecteplase treatment group
Drug: alteplase — alteplase
  Arms: Alteplase active control group

SUMMARY:
This study is open to Chinese adults who had an ischaemic stroke, which means that blood vessels in the brain are blocked. To resolve blood clots, people in the study get either tenecteplase or alteplase within 4 hours and 30 minutes after stroke. The purpose of this study is to compare how tenecteplase and alteplase improve peoples' recovering of physical activity. Alteplase is standard of care. Tenecteplase is a modified variant of alteplase that is easier to administer and is approved to treat heart attack. This study is to find out whether tenecteplase is as good as alteplase in people with ischaemic stroke.

Participants are equally put into 2 treatment groups by chance. Participants in one group get tenecteplase as a single injection into a vein. Participants in the other group get alteplase as an injection into a vein (10% of the dose) and the remainder as an infusion over 1 hour.

Participants are in the study for about 3 months. They are in the hospital for the first week after treatment. Then they visit the study site 1 and 3 months after treatment. At these visits, peoples' ability to independently carry out daily activities is assessed. Scores for physical activity are compared between both treatment groups. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of ischaemic stroke with a measurable neurological deficit on National Institutes of Health Stroke Scale (NIHSS) (0< NIHSS ≤25); if NIHSS <4, patients have to be with at least a measurable deficit on motor power (upper or lower limbs ≥1)
* Stroke symptoms should have been present for at least 30 minutes (min) without significant improvement prior to randomisation
* Thrombolytic therapy can be initiated within 4.5 Hour(s) (h) of Acute ischaemic stroke (AIS) onset
* Patients with premorbid modified Rankin Scale (mRS) 0 or 1
* Signed and dated written informed consent in accordance with good clinical practice (GCP) and local legislation prior to trial admission

Exclusion Criteria:

* Evidence of intracranial haemorrhage on the Computed tomography (CT) scan or symptoms suggestive of subarachnoid haemorrhage, even if the CT scan is normal
* Patients who must or are expected to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Acute bleeding diathesis, including but not limited to

  * Known genetic predisposition to bleeding or significant bleeding disorder at present or within the past 6 Month(s) (m)
  * Administration of heparin within the previous 48 h and activated partial thromboplastin time (aPTT) exceeding the upper limit of normal for laboratory measurement
  * Current use of vitamin K based oral anticoagulants (e.g. warfarin) and a prolonged prothrombin time (International normalised Ratio (INR) > 1.7 or Prothrombin time (PT)>15 seconds (s)) or current use of novel oral anticoagulants (i.e. dabigitran, rivaroxiban, or apixiban) with prolongation of activated partial thromboplastin time (aPTT) and/or PT above the upper limit of the local laboratory reference range
  * Platelet count of below 100,000/mm3 at screening
  * Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
  * Recent traumatic external heart massage, obstetrical delivery, or recent puncture of a non-compressive blood-vessel (e.g. subclavian or jugular vein puncture) , within the past 10 days
  * Known history of suspected intracranial haemorrhage or suspected subarachnoid haemorrhage from aneurysm
  * Neoplasm with increased haemorrhagic risk
  * Documented ulcerative gastrointestinal disease during the last 3 m, oesophageal varices, arterial aneurysm, or arterial/venous malformations
  * Any known disorder associated with a significant increased risk of bleeding
* Bacterial endocarditis or pericarditis at screening
* Acute pancreatitis at screening
* Significant trauma or major surgery (according to the investigator's assessment) in the past 3 m
* Imaging demonstrates multi-lobar infarction (hypodensity >1/3 cerebral hemisphere)
* Severe uncontrolled arterial hypertension, e.g. systolic blood pressure (BP) >185 mmHg or diastolic BP >110 mmHg Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1489 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- China (55):
  - Inner Mongolia Baogang Hospital, Baotou
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Beijing Tiantan Hospital affiliated to Cap Med University, Beijing
  - Beijing Tongren Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The third xiangya hospital of Central South University, Changsha
  - Hexigten Banner Mongolian Traditional Chinese medicine hospital, Chifeng
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Center Hospital of Dalian, Dalian
  - Daqing People's Hospital, Daqing
  - Shengli Oilfield central hospital, Dongying
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Huai'an Second People's Hospital, Huai'an
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia
  - The second Hospital of Jiaxing, Jiaxing
  - Center Hospital of Jinan, Jinan
  - Jinhua Municipal Central Hospital, Jinhua
  - The first People's Hospital of Lianyungang, Lianyungang
  - Linfen Central Hospital, Linfen
  - Linyi People's Hospital, Linyi
  - The First People's Hospital of Tancheng County, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The First People's Hospital of Nanning, Nanning
  - The First People's Hospital of Nantong, Nantong
  - Ruian People's Hospital, Ruian
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai Seventh People's Hospital, Shanghai
  - Affiliated Central Hospital of Shenyang Medical College, Shenyang
  - The First People's Hospital of Shenyang, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - The 2nd Hospital of Tianjin Medical University, Tianjin
  - The First Center Hospital of Tianjin, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Xianyang Hospital of Yan'an University, Xianyang
  - Xinxiang Central Hospital, Xinxiang
  - The People's Hospital Of Xuancheng City, Xuancheng
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Affiliated Hospital of Yangzhou University, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Yiyang Central Hospital, Yiyang

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Meng X, Li S, Dai H, Lu G, Wang W, Che F, Geng Y, Sun M, Li X, Wang Y. Tenecteplase Versus Alteplase in Acute Ischemic Stroke in Chinese Patients: Protocol for the ORIGINAL Study. Stroke Vasc Interv Neurol. 2024 May 7;4(4):e001363. doi: 10.1161/SVIN.124.001363. eCollection 2024 Jul. PMID 41585404
- [Derived] Meng X, Li S, Dai H, Lu G, Wang W, Che F, Geng Y, Sun M, Li X, Li H, Wang Y. Tenecteplase vs Alteplase for Patients With Acute Ischemic Stroke: The ORIGINAL Randomized Clinical Trial. JAMA. 2024 Nov 5;332(17):1437-1445. doi: 10.1001/jama.2024.14721. PMID 39264623
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main objective of this multi-centre, prospective, randomised, open label, blinded endpoint (PROBE), active-controlled parallel group phase III trial was to assess whether tenecteplase was non-inferior to alteplase in favourable outcome in Chinese patients with acute ischaemic stroke (AIS) who were eligible for intravenous (i.v.) thrombolysis within 4.5 h of symptom onset.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Tenecteplase Treatment Group: Chinese patients with AIS were screened (visit 1) and randomised (visit 2a) when admitted. Patients received a single dose of tenecteplase, 0.25 mg/kg via intravenous (iv) bolus no later than 4.5 hours (h) after symptom onset. Visits on Day 1 consisted of two further visits (Visit 2b and Visit 2c) that were performed 1 h and 2 h after the start of the treatment. Visits 3 to 5 for continuous follow-up were performed on day 2, 8 and 30 after the start of the treatment. Treated patients performed a 90-day follow-up visit after the treatment to complete the study.
- Alteplase Active Control Group: Chinese patients with AIS were screened (visit 1) and randomised (visit 2a) when admitted. Patients received a single dose of alteplase, 0.9 mg/kg, 10% via intravenous (iv) bolus and the remaining 90% of the total dose administered as an iv infusion over 1 h no later than 4.5 hours (h) after symptom onset. Visits on Day 1 consisted of two further visits (Visit 2b and Visit 2c) that were performed 1 h and 2 h after the start of the treatment. Visits 3 to 5 for continuous follow-up were performed on day 2, 8 and 30 after the start of the treatment. Treated patients performed a 90-day follow-up visit after the treatment to complete the study.
Period: Overall Study
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Started | 744 | 745
Treated | 733 | 735
Completed | 671 | 675
Not Completed | 73 | 70
Not completed — Lost to Follow-up | 20 | 10
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Death | 34 | 44
Not completed — not treated | 3 | 6
Not completed — Investigator removed subject | 1 | 2
Not completed — questionnaire result not evaluated | 1 | 0
Not completed — refuse of hospital visit | 1 | 3
Not completed — Subject withdrew | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): This patient set included all randomised patients who received any dose of treatment. Treatment assignment was as randomised. This was the primary analysis set for presentation of efficacy according to the intention-to-treat principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group | Total
Number analyzed (Participants) | 732 | 733 | 1465
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (11.1) | 65.0 (11.1) | 65.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 231 | 446
  Male | 517 | 502 | 1019
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 732 | 733 | 1465
  Unknown or Not Reported | 0 | 0 | 0
National Institutes of Health Stroke Scale (NIHSS) class 1 at baseline [Count of Participants; unit: Participants] — Total NIHSS score (0-42) = sum of 11 individual item scores, higher total scores meaning more severe deficits.
  individual domains: level of consciousness (LOC), best gaze, visual fields, facial paresis, motor function arms, motor function legs, limb ataxia, sensory, language, dysarthria, extinction and inattention.
  Mild strokes (NIHSS < 6): High likelihood of good recovery and independence, Moderate strokes (NIHSS 6-15): Variable outcomes depending on timely intervention, Severe strokes (NIHSS > 15): Lower likelihood of recovery without significant disability and higher risk of mortality.
  Participants
    NIHSS total score <6 | 299 | 297 | 596
    NIHSS total score 6 - 15 | 390 | 393 | 783
    NIHSS total score >=15 | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Score of 0 or 1
Description: Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death). It was measured at Day 90.
  Percentages are rounded to the nearest digits.
Time Frame: At Day 90±7 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 733
Percentage of participants | 72.7 | 70.3
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Non-Inferiority — pre-specified non-inferiority margin for risk ratio = 0.937; Modified Possion Regression Model; treatment = main effect; baseline NHISS, age + time to drug administration since stroke symptoms onset = continuous covariates; Risk Ratio (RR) = 1.0278, 95% CI 2-sided [0.9678 to 1.0915] — tenecteplase versus alteplase

2. Secondary Outcome: Percentage of Participants With Major Neurological Improvement (National Institutes of Health Stroke Scale (NIHSS) Score of 0 or Improvement of at Least 4 Points Compared With Baseline
Description: Total NIHSS score (0-42) = sum of 11 individual item scores, higher total scores meaning more severe deficits.
  indivudal domains: level of consciousness (LOC), best gaze, visual fields, facial paresis, motor function arms, motor function legs, limb ataxia, sensory, language, dysarthria, extinction and inattention.
  Mild strokes (NIHSS < 6): High likelihood of good recovery and independence, Moderate strokes (NIHSS 6-15): Variable outcomes depending on timely intervention, Severe strokes (NIHSS > 15): Lower likelihood of recovery without significant disability and higher risk of mortality.
  Percentages are rounded to the nearest digits.
Time Frame: At 24 hours
Population: Full Analysis Set (FAS), This endpoint analysis is based on observed cases, no imputation performed for patients missing NIHSS score at 24h.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 711 | 716
Percentage of participants | 48.0 | 45.0
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other — log-binomial regression model; p = 0.2412, Regression, Linear — p-value was for superiority testing; treatment = main effect; baseline NHISS, age + time to drug administration since stroke symptoms onset = covariates; Risk Ratio (RR) = 1.0671, 95% CI 2-sided [0.9573 to 1.1895] — tenecteplase versus alteplase

3. Secondary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Score of 0-2
Description: Percentage of participants with Modified Rankin Scale (mRS) score of 0-2 is presented.
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death). It was measured at Day 90.
  Percentages are rounded to the nearest digits.
Time Frame: At Day 90
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 733
Percentage of participants | 80.9 | 79.9
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other — Modified Poisson regression model; p = 0.7480, Regression, Linear — p-value was for superiority testing; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.0078, 95% CI 2-sided [0.9614 to 1.0564] — tenecteplase versus alteplase

4. Secondary Outcome: Change From Baseline of National Institutes of Health Stroke Scale (NIHSS) Score
Description: Total NIHSS score (0-42) = sum of 11 individual item scores, higher total scores meaning more severe deficits.
  indivudal domains: level of consciousness (LOC), best gaze, visual fields, facial paresis, motor function arms, motor function legs, limb ataxia, sensory, language, dysarthria, extinction and inattention.
  Restricted maximum likelihood (REML) based MMRM approach used to compare change from baseline in NIHSS score at day 90. If patient misses visit, missing data will not be imputed. The mixed effect model will handle missing data based on a likelihood method under MAR assumption.
  Change in NIHSS score from baseline = overall mean + treatment + visit + baseline NIHSS + age + time to drug administration since onset of stroke symptoms + treatment by visit interaction + baseline NIHSS by visit interaction + random error.
Time Frame: At baseline and at Day 90
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 733
score on a scale | -3.47 (0.34) | -3.02 (0.34)
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other; p = 0.3511, Mixed Models Analysis; baseline NIHSS, age, time to administration since stroke symptoms onset = linear covariates; treatment = fixed effects; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.40 to 0.50], Standard Error of Mean 0.48 — Difference in LSmean tenecteplase vs alteplase

5. Secondary Outcome: Distribution of Modified Rankin Scale (mRS)
Description: Distribution of Modified Rankin Scale (mRS) is presented. Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death). It was measured at Day 90.
Time Frame: At Day 90
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 733
Percentage of participants
  mRS score = 0 | 40.3 | 40.5
  mRS score = 1 | 30.1 | 28.2
  mRS score = 2 | 7.8 | 9.4
  mRS score = 3 | 6.7 | 5.5
  mRS score = 4 | 4.8 | 6.4
  mRS score = 5 | 1.9 | 1.6
  mRS score = 6 | 4.6 | 6.0
  missing | 3.8 | 2.3
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other; p = 0.4806, Regression, Logistic; Assumption-free ordinal analysis; Odds Ratio (OR) = 1.0418 — tenecteplase versus alteplase

6. Secondary Outcome: Percentage of Participants With Barthel Index Score ≥95
Description: The Barthel Index is an ordinal scale used to measure performance in activities of daily living (ADL). The Barthel Index consists of 10 items. The total score of the Barthel Index ranges from 0 to 100, and higher scores indicate better outcome.
  Percentages are rounded to the nearest digits.
Time Frame: up to 90 days
Population: Full Analysis Set (FAS), No imputation was performed on patients missing Bathel Score at day 90.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 699 | 708
Percentage of participants | 75.7 | 73.9
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other — Poisson regression model; p = 0.5116, Regression, Linear; treatment = main effect; baseline NHISS, age + time to drug administration since stroke symptoms onset = covariates; Risk Ratio (RR) = 1.0189, 95% CI 2-sided [0.9635 to 1.0774] — tenecteplase versus alteplase

7. Secondary Outcome: Percentage of Participants With Symptomatic Intracerebral Haemorrhage (sICH) Per European Cooperative Acute Stroke Study (ECASS) Ⅲ Definition During On-treatment Period
Description: Percentage of participants with Symptomatic Intracerebral Haemorrhage (sICH) per European Cooperative Acute Stroke Study (ECASS) Ⅲ definition during on-treatment period is presented.
  Percentages are rounded to the nearest digits.
Time Frame: Up to 7 days.
Population: Safety set (SS): This patient set included all patients who were randomised and received any dose of treatment. It was the main analysis set for presentation of safety. Patients were analysed according to the actual treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 736
Percentage of participants | 1.2 | 1.2
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other; p = 1.000, Suissa-Shuster test; Risk Ratio (RR) = 1.005, 95% CI 2-sided [0.370 to 2.701] — tenecteplase versus alteplase

8. Secondary Outcome: Percentage of Participants Who Died by Day 90
Description: Percentage of participants who died by day 90 is presented. Percentages are rounded to the nearest digits.
Time Frame: up to 90 days
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 736
Percentage of participants | 4.6 | 5.8
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other; p = 0.303, Chi-squared; Risk Ratio (RR) = 0.795, 95% CI 2-sided [0.513 to 1.232] — tenecteplase versus alteplase

9. Secondary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Score of 5 or 6
Description: Percentage of participants with Modified Rankin Scale (mRS) score of 5 or 6 is presented.
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death). It was measured at Day 90.
  Percentages are rounded to the nearest digits.
Time Frame: At Day 90
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase Treatment Group | Alteplase Active Control Group
Number analyzed (Participants) | 732 | 733
Percentage of participants | 6.8 | 7.8
Statistical Analysis 1: Comparison: Tenecteplase Treatment Group vs Alteplase Active Control Group; Test type: Other — Modified Poisson regression model; p = 0.6345, Regression, Linear — p-value was for superiority testing; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.9215, 95% CI 2-sided [0.6578 to 1.2908] — tenecteplase versus alteplase

ADVERSE EVENTS:
Time Frame: AEs are reported for the on-treatment period from start of treatment until end of residual effect period, up to 7 days. All cause mortality was reported from start of treatment until death by any cause, up to 97 days.
Description: Safety set (SS): This patient set included all patients who were randomised and received any dose of treatment. It was the main analysis set for presentation of safety. Patients were analysed according to the actual treatment.
Arm/Group | Alteplase Active Control Group | Tenecteplase Treatment Group
All-Cause Mortality (participants affected / at risk) | 44/736 | 34/732
Serious Adverse Events (participants affected / at risk) | 115/736 | 116/732
Other Adverse Events (participants affected / at risk) | 347/736 | 334/732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase Active Control Group (N=736) | Tenecteplase Treatment Group (N=732)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 8 | 8
Cardiac failure acute (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial injury (Cardiac disorders) | 1 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Stress ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Condition aggravated (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Encephalitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Intracranial infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 7
Pneumonia aspiration (Infections and infestations) | 6 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 8 | 7
Spleen contusion (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 4 | 6
Brain oedema (Nervous system disorders) | 4 | 6
Brain stem haemorrhage (Nervous system disorders) | 3 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Carotid artery dissection (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 3 | 0
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 2 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 21 | 25
Cerebral infarction (Nervous system disorders) | 14 | 16
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 4 | 0
Decorticate posture (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 3 | 2
Haemorrhage intracranial (Nervous system disorders) | 7 | 5
Haemorrhagic cerebral infarction (Nervous system disorders) | 7 | 3
Haemorrhagic transformation stroke (Nervous system disorders) | 16 | 10
Hemiparesis (Nervous system disorders) | 0 | 3
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 5
Thalamus haemorrhage (Nervous system disorders) | 1 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Delirium (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Aortic dissection (Vascular disorders) | 1 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 13 | 8
Embolism venous (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 1 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase Active Control Group (N=736) | Tenecteplase Treatment Group (N=732)
Anaemia (Blood and lymphatic system disorders) | 37 | 32
Constipation (Gastrointestinal disorders) | 123 | 131
Gingival bleeding (Gastrointestinal disorders) | 78 | 79
Pyrexia (General disorders) | 43 | 33
Pneumonia (Infections and infestations) | 65 | 55
Urinary tract infection (Infections and infestations) | 49 | 44
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 45 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 77 | 70
Hypoproteinaemia (Metabolism and nutrition disorders) | 41 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04915729/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT04915729/SAP_001.pdf